CLINICAL TRIAL: NCT01755624
Title: A Phase II Randomized Study of TTField Therapy (150 kHz) Versus Supportive Care in Non-small Cell Lung Cancer Patients With 1-5 Brain Metastases Following Optimal Standard Local Treatment
Brief Title: Effect of TTFields (150kHz) in Non-small Cell Lung Cancer (NSCLC) Patients With 1-5 Brain Metastases Following Optimal Standard Local Treatment (COMET)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF-21
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-07

CONDITIONS: 1-5 Brain Metastases From Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Brain metastases; Treatment; Minimal toxicity; TTFields; TTF; Tumor Treating Fields; NovoCure
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NovoTTF-100A device (Experimental): Patients will be treated continuously with the NovoTTF-100A device. NovoTTF-100A treatment will consist of wearing four electrically insulated electrode arrays on the head. The treatment enables the patient to maintain regular daily routine.
  Interventions: Device: NovoTTF-100A device
- Best Standard of Care (Active Comparator): Patients will be treated as the best known standard of care for Non-Small Cell Lung Cancer metastatic to the brain.
  Interventions: Other: Best Standard of Care

INTERVENTIONS:
Device: NovoTTF-100A device
  Arms: NovoTTF-100A device
Other: Best Standard of Care
  Arms: Best Standard of Care

SUMMARY:
The study is a prospective, randomly controlled phase II trial, designed to test the efficacy, safety and neurocognitive outcomes of a medical device, the NovoTTF-100A, in the treatment of NSCLC patients with controlled systemic disease, following optimal standard local treatment for 1-5 brain metastases (BM). The device is an experimental, portable, battery operated device for chronic administration of alternating electric fields (termed TTFields or TTF) to the region of the malignant tumor, by means of surface, insulated electrode arrays.

DETAILED DESCRIPTION:
PAST PRE CLINICAL AND CLINICAL EXPERIENCE:

The effect of the electric fields generated by the NovoTTF-100A device (TTFields, TTF) has demonstrated significant activity in in vitro and in vivo NSCLC pre-clinical models both as a single modality treatment and in combination with chemotherapies. TTField therapy has also shown to inhibit metastatic spread of malignant melanoma in in vivo experiment.

In a small scale pilot study, patients with stage IIIB- IV NSCLC who had had tumor progression after at least one line of prior chemotherapy received Pemetrexed together with TTField therapy applied to the chest and upper abdomen until disease progression. Efficacy endpoints were remarkably high compared to historical data for Pemetrexed alone.

In a large prospective, randomized trial, in recurrent GBM. The outcome of subjects treated with the NovoTTF-100A device was compared to those treated with an effective best standard of care chemotherapy (including bevacizumab). NovoTTF-100A subjects had comparable overall survival to subjects receiving the best available chemotherapy in the US today. Similar results showing comparability of NovoTTF-100A to BSC chemotherapy were seen in all secondary endpoints. Recurrent GBM patients treated with the NovoTTF-100A device in this trial experienced fewer side effects in general, significantly fewer treatment related side effects, and significantly lower gastrointestinal, hematological and infectious adverse events compared to controls. The only device-related adverse events seen were a mild to moderate skin irritation beneath the device electrodes. Finally, quality of life measures were better in NovoTTF-100A subjects as a group when compared to subjects receiving effective best standard of care chemotherapy.

DESCRIPTION OF THE TRIAL:

All patients included in this trial are diagnosed with NSCLC, and have stable systemic disease with 1-5 supratentorial brain metastases who are amenable to optimal standard local treatment (surgical resection/stereotactic radio surgery (SRS)/both). In addition, all patients must meet all eligibility criteria.

Eligible patients will be randomly assigned to one of two groups:

1. Treatment with the NovoTTF-100A device together with best standard of care.
2. Best standard of care

Patients will be randomized at a 1:1 ratio. Baseline tests will be performed in patients enrolled in both arms. If assigned to the NovoTTF-100A group, the patients will be treated continuously with the device until disease progression in the brain.

On both arms, patients who recur in the brain will be offered one of the following salvage treatments (according to local practice) including, but not limited to:

1. Surgery (or repeat surgery)
2. SRS (or repeat SRS)
3. Whole brain radiotherapy (WBRT)

Patients on Arm II may cross over to TTFields therapy after salvage therapy if investigators believe it is in the best interest of the patients and patients agree.

NovoTTF-100A treatment will consist of wearing four electrically insulated electrode arrays on the head. Electrode array placement will require shaving of the scalp before and frequently during the treatment. After an initial short visit to the clinic for training and monitoring, patients will be released to continue treatment at home where they can maintain their regular daily routine.

During the trial, regardless of which treatment group the patient was assigned to, he or she will need to return once every month to the clinic where an examination by a physician and a routine laboratory examinations will be done. These routine visits will continue for as long as the patient's disease is not progressing in the brain.

During the monthly follow up visits to the clinic patients will be examined physically and neurologically. Additionally, routine blood tests will be performed. A routine MRI of the head will be performed at baseline and every third month thereafter, until disease progression in the brain. In addition a neurocognitive test will be performed at baseline and every third month thereafter, until disease progression in the brain. After this follow up plan, patients will be contacted once per month by telephone to answer basic questions about their health status.

SCIENTIFIC BACKGROUND:

Electric fields exert forces on electric charges similar to the way a magnet exerts forces on metallic particles within a magnetic field. These forces cause movement and rotation of electrically charged biological building blocks, much like the alignment of metallic particles seen along the lines of force radiating outwards from a magnet.

Electric fields can also cause muscles to twitch and if strong enough may heat tissues. TTFields are alternating electric fields of low intensity. This means that they change their direction repetitively many times a second. Since they change direction very rapidly (150 thousand times a second), they do not cause muscles to twitch, nor do they have any effects on other electrically activated tissues in the body (brain, nerves and heart). Since the intensities of TTFields in the body are very low, they do not cause heating.

The breakthrough finding made by Novocure was that finely tuned alternating fields of very low intensity, now termed TTFields (Tumor Treating Fields), cause a significant slowing in the growth of cancer cells. Due to the unique geometric shape of cancer cells when they are multiplying, TTFields cause the building blocks of these cells to move and pile up in such a way that the cells physically explode. In addition, cancer cells also contain miniature building blocks which act as tiny motors in moving essential parts of the cells from place to place. TTFields cause these tiny motors to fall apart since they have a special type of electric charge.

As a result of these two effects, cancer tumor growth is slowed and can even reverse after continuous exposure to TTFields.

Other cells in the body (normal healthy tissues) are affected much less than cancer cells since they multiply at a much slower rate if at all. In addition TTFields can be directed to a certain part of the body, leaving sensitive areas out of their reach.

In conclusion, TTField hold the promise of serving as a brand new cancer treatment with very few side effects and promising affectivity in slowing or reversing this disease.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older
2. Life expectancy of ≥ 3 months
3. Performance status WHO 0-2 (may be assessed under steroid therapy)
4. New diagnosis of BM from a histologically or cytologically confirmed primary or metastatic NSCLC tumor, meeting 1 of the following criteria:

   1. Stable systemic cancer for the last 3 months (achieved by surgery, radiotherapy, or chemotherapy), defined as absence of symptomatic and radiological progression, according to RECIST Criteria
   2. Asymptomatic synchronous primary tumor (treatable by surgery, radiotherapy, or chemotherapy)
5. BM biopsy required if no extracranial tumor (unknown primary tumor) OR extracranial diagnosis made more than 4 years previously
6. Must have one to five brain lesions, confirmed by contrast enhanced MRI, all amenable either surgical resection, or to SRS according to the following criteria:

   1. Largest diameter ≤ 3.5 cm for single metastasis
   2. Largest diameter ≤ 2.5 cm for 2 to 5 metastases
7. Stable or decreasing dose of steroids for at least 5 days before screening
8. Patients must be receiving optimal therapy for their extracranial disease according to local practice at each center. Patients may continue on systemic therapy while receiving TTField therapy

Exclusion Criteria:

1. Infratentorial metastases
2. Leptomeningeal metastases
3. Patients who previously received WBRT or SRS for BM (prior resection is allowed as long as any remaining tumor is treated under the protocol)
4. Significant co-morbidity which is expected to affect patient's prognosis or ability to receive optimal systemic therapy:

   1. Inadequate and clinically relevant hematological, hepatic and renal abnormalities defined as: Neutrophil count > 1.5 x 10 9/L and platelet count > 100 x 10 9/L; bilirubin < 1.5 x ULN; AST and/or ALT < 2.5 x ULN or < 5 x ULN is patient has documented liver metastases; and serum creatinine < 1.5 x ULN
   2. History of significant cardiovascular disease unless the disease is well controlled. Significant cardiac disease includes second/third degree heart block; significant ischemic heart disease; poorly controlled hypertension; congestive heart failure of the New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary activity results in fatigue, palpitation or dyspnea).
   3. History of arrhythmia that is symptomatic or requires treatment. Patients with atrial fibrillation or flutter controlled by medication are not excluded from participation in the trial
   4. History of cerebrovascular accident (CVA) within 6 months prior to randomization
   5. Active infection or serious underlying medical condition that would impair the ability of the patient to received protocol therapy
   6. History of any psychiatric condition that might impair the patient's ability to understand or comply with the requirements of the study or to provide consent
   7. Pregnant, or women with an intact uterus (unless amenorrhoeic for the last 24 months) not using effective means of contraception
5. Unable to operate the NovoTTF-100A device independently or with the help of a caregiver
6. Implantable electronic medical devices in the brain
7. Known allergies to medical adhesives or hydrogel
8. Concurrent brain directed therapy (beyond SRS, surgery and TTField therapy as per protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Time to Local and Distant Progression in The Brain | 2 years

SECONDARY OUTCOMES:
Overall Survival | 2 years
6-Month Disease Control Rate in The Brain | 2 years
Neurocognitive Function (MMSE and HVLT) | 2 years
Quality of life (QLQ-C30 and BN-20) | 2 years
Overall (systemic) Progression-Free Survival (RECIST Criteria) | 2 years
Adverse Events Severity and Frequency | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Salamaggi, MD, Principal Investigator — Lecco General Hospital
Locations (7):
- Na Homolce Hospital, Prague, Czechia
- France (2):
  - Hopital Neurologique Pierre Wertheimer, Lyon
  - Centre Paul Strauss, Strasbourg
- Ospedale Lecco, Lecco, Italy
- Poland (2):
  - Medical University of Gdańsk, Gdansk
  - Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
- ICO L'Hospitalet - Hospital Duran i Reynals, Barcelona, Spain

REFERENCES:
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Kirson ED, Giladi M, Gurvich Z, Itzhaki A, Mordechovich D, Schneiderman RS, Wasserman Y, Ryffel B, Goldsher D, Palti Y. Alternating electric fields (TTFields) inhibit metastatic spread of solid tumors to the lungs. Clin Exp Metastasis. 2009;26(7):633-40. doi: 10.1007/s10585-009-9262-y. Epub 2009 Apr 23. PMID 19387848
- [Background] Pless M, Weinberg U. Tumor treating fields: concept, evidence and future. Expert Opin Investig Drugs. 2011 Aug;20(8):1099-106. doi: 10.1517/13543784.2011.583236. Epub 2011 May 9. PMID 21548832
- [Background] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Background] Pless M, Droege C, von Moos R, Salzberg M, Betticher D. A phase I/II trial of Tumor Treating Fields (TTFields) therapy in combination with pemetrexed for advanced non-small cell lung cancer. Lung Cancer. 2013 Sep;81(3):445-450. doi: 10.1016/j.lungcan.2013.06.025. Epub 2013 Jul 23. PMID 23891283
- [Background] Weinberg, U., et al. An Open Label Pilot Study of Tumor Treating Fields (TTFields) in Combination with Pemetrexed for Advanced Non-small Cell Lung Cancer (NSCLC). in ERS Annual Congress. 2010. Publisher: Abstract 363.